CLINICAL TRIAL: NCT01113476
Title: Phase I Study of Combination of Nab-paclitaxel, Gemcitabine, and Bevacizumab in Advanced Malignancies
Brief Title: Nab-paclitaxel, Gemcitabine, and Bevacizumab in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0855; NCI-2011-02061 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Malignancies; Nab-paclitaxel; Gemcitabine; Bevacizumab
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Paclitaxel; Albumin-Bound Paclitaxel; Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel, Gemcitabine + Bevacizumab (Experimental): Starting doses of Nab-paclitaxel 50 mg/m^2, Bevacizumab 5 mg/kg + fixed dose of Gemcitabine 1000 mg/m^2
  Interventions: Drug: Nab-paclitaxel; Drug: Bevacizumab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel — Starting dose of 50 mg/m^2 on Day 1, 8 + 15 every 28 days (+/- 2 days)
  Other Names: Paclitaxel; Abraxane; ABI-007
Drug: Bevacizumab — Starting dose of 5 mg/m^2 on Day 1 + 15 every 28 days (+/- 2 days)
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Gemcitabine — 1000 mg/kg Day 1, 8 + 15 every 28 days (+/- 2 days)
  Other Names: Gemcitabine Hydrochloride; Gemzar

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Abraxane (nab-paclitaxel), Gemzar (gemcitabine), and Avastin (bevacizumab) that can be given to patients with advanced cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of a combination of nab-paclitaxel, gemcitabine, and bevacizumab based on when you joined this study. All participants will receive the same dose level of gemcitabine. However, the first group of participants will receive the lowest dose level of nab-paclitaxel and bevacizumab. Each new group will receive a higher dose for one of the drugs than the group before it, if no intolerable side effects were seen. The other drug may be at the same dose or a lower dose. This will continue until the highest tolerable dose of combination of nab-paclitaxel, gemcitabine, and bevacizumab is found. Up to 15 dose levels of the study drug combination will be tested. Three (3) to 4 participants will be enrolled at each dose level.

Once the highest tolerated dose is found, up to 10 more participants will be added at that dose level. This is called an expansion group.

Study Drug Administration:

On Days 1, 8, and 15 of each 28-day cycle, you will receive nab-paclitaxel and gemcitabine by vein over about 90 minutes total. Also, if the first dose is well tolerated, you may be given the remaining doses of nab-paclitaxel and gemcitabine at home.

On Days 1 and 15 of each cycle, you will receive bevacizumab by vein over about 60 minutes. Also, if the first dose is well tolerated, you may be given the remaining doses of bevacizumab at home.

Study Visits:

Each week during Cycle 1:

* Your medical history will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* Blood (about 2-5 teaspoons) will be drawn to test for fat levels in the blood. You will need to fast for at least 4 hours before this blood draw.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.
* You will have urine tests performed to check for high levels of protein in your urine (a known side effect of bevacizumab).

On Day 1 and 8 of Cycle 1, you will have a physical exam, including measurement of your weight and vital signs.

During Week 1 of Cycles 2 and beyond:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* Blood (about 2-5 teaspoons) will be drawn to test for fat levels in the blood. You will need to fast for at least 4 hours before this blood draw.
* Blood (about 2 teaspoons) will be drawn to see how well your blood clots and how long it takes for your blood to clot.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.
* Females who are able to become pregnant must have a negative blood (about 1 teaspoon) pregnancy test.

During Weeks 2 and 4 of Cycles 2 and beyond:

* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.
* Blood (about 2 teaspoons) will be collected for routine tests.

During Week 3 of Cycles 2 and beyond:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* Blood (about 2-5 teaspoons) will be drawn to test for fat levels in the blood. You will need to fast for at least 4 hours before this blood draw.
* Blood (about 2 teaspoons) will be drawn to see how well your blood clots and how long it takes for your blood to clot.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on), you will have an x-ray, CT scan, PET scan, or MRI scan to check the status of the disease. If you have disease in your bones, a bone scan may also be done.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

You may chose to stop taking the study drugs at any time. You should tell the study doctor right away if you are thinking about stopping your participation in this study. The study doctor will talk to you about how to safely stop taking the study drugs.

This is an investigational study. Gemcitabine is FDA approved and commercially available for the treatment of certain types of breast cancer, non-small cell lung cancer, pancreatic cancer, and ovarian cancer. Bevacizumab is FDA approved and commercially available for the treatment of colorectal, breast, lung, and brain cancer. Nab-paclitaxel is FDA approved and commercially available for the treatment of breast cancer. The combination of these drugs is investigational.

Up to 120 patients will take part in this study, but this may be increased at a later time. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that induces a CR rate of at least 10% or improves survival by at least three months.
2. Patients should be at least four weeks from the last day of therapeutic radiation or cytotoxic chemotherapy or from antibody therapy, or at least five half-lives from non-cytotoxic targeted or biologic therapy. Patients may have received palliative radiation immediately before (or during) treatment provided radiation is not to the only target lesion available.
3. ECOG performance status </= 2 (Karnofsky >/= 60%).
4. Patients must have allowable organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/=50,000/mL; creatinine </= 3 X ULN; total bilirubin </= 3.0; ALT(SGPT) </= 5 X ULN; fasting level of total cholesterol of no more than 350mg/dL; triglyceride level of no more than 400mg/dL.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Patients may not be receiving any other investigational agents and/or any other concurrent anticancer agents or therapies.

Exclusion Criteria:

1. Patients with hemoptysis within 28 days prior to entering the study.
2. Patients with clinically significant unexplained bleeding within 28 days prior to entering the study.
3. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140mmHg, diastolic blood pressure > 90 mmHg on medication).
4. Pregnant or lactating women.
5. History of hypersensitivity to bevacizumab, murine products, or any component of the formulation.
6. History of hypersensitivity to gemcitabine.
7. History of hypersensitivity to nab-paclitaxel or paclitaxel.
8. Patients with clinically significant cardiovascular disease: Myocardial Infarction or unstable angina pectoris within the last 6 months, Class III/IV NYHA heart failure.
9. History of CVA within 6 months.
10. History of surgery within last 28 days.
11. Grade 3/4 proteinuria.
12. Nephrotic syndrome.
13. Incompletely healed wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Gemcitabine, Nab-Paclitaxel and Bevacizumab | With each 28 day cycle
  A MTD is defined as the dose level below the dose at which 2 of 6 patients experience drug-related dose limiting toxicity (DLT) in the first cycle. DLT defined as any grade 3 or 4 non-hematologic toxicity as defined in the NCI CTC v4.0, even if expected and believed related to study medications (except nausea and vomiting responsive to appropriate regimens or alopecia), any Grade 4 hematologic toxicity lasting 2 weeks or longer (as defined by the NCI-CTCAE), despite supportive care; any Grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other Grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in the NCI-CTCAE v.4.0 that is attributable to therapy.

SECONDARY OUTCOMES:
Response Rate | After 2, 28 day cycles
  Patients with lymphoma measured per WHO criteria, all others evaluated with RECIST (version 1.1) criteria. Measurable disease defined as at least one lesion that can be accurately measured in at least one dimension. Best Response: Measurement of longest dimension of each lesion size is required for follow-up. Complete Response (CR): Disappearance of all target and non-target lesions and no evidence of new lesions documented by 2 disease assessments at least 4 weeks apart. Partial Response (PR): At least 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions, taking as reference baseline sum of LD. Stable Disease (SD): Stable disease defined as any condition not meeting above criteria. Progressive Disease (PD): At least a 20% increase in sum of LD of target lesions taking as reference smallest sum LD or appearance of new lesions after study entry.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sen S, Kato S, Agarwal R, Piha-Paul S, Hess K, Karp D, Janku F, Fu S, Naing A, Pant S, Falchook G, Tang C, Wu X, Ye Y, Tsimberidou A, Subbiah V, Kurzrock R, Byers L, Westin S, Lim J, Bean S, Bass A, Nguyen L, Meric-Bernstam F, Hong D. Phase I study of nab-paclitaxel, gemcitabine, and bevacizumab in patients with advanced cancers. Br J Cancer. 2018 May;118(11):1419-1424. doi: 10.1038/s41416-018-0068-z. Epub 2018 Apr 26. PMID 29695765
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org